CLINICAL TRIAL: NCT05511961
Title: Ameliorating Child Poverty Through Connecting Economic Services With Child Health Services (ACCESS): A Randomised Controlled Trial of the Healthier Wealthier Families Model in Sweden
Brief Title: A Randomised Controlled Trial of Healthier Wealthier Families in Sweden
Acronym: ACCESS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Full trial considered unfeasible after internal pilot. Internal pilot to be published. Record will be updated when publication available.
Sponsor: Uppsala University (Other)
Responsible Party: Principal Investigator, Anna Sarkadi, Professor, Uppsala University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2021-01415
Record Dates: First submitted 2022-08-19; First posted 2022-08-23 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-04

CONDITIONS: Material and Social Deprivation: An Enforced Lack of Necessary and Desirable Items to Lead an Adequate Life
Keywords: Child poverty, Economic services, Child health services; Healthier Wealthier Families, Sweden

STUDY DESIGN:
Intervention Model Description: A two-arm randomised waitlist-control superiority trial (1:1 allocation ratio) will be conducted to evaluate the effectiveness of the HWF model in improving the financial situation of families who have self-reported economic difficulties. The intervention arm will be referred to budget and debt counselling immediately after randomisation and the waitlist-control arm around 3 months later. Both arms will be offered a financial guidance book at randomisation. Randomised controlled trial (RCT) assessments will take place at two points: pre-intervention (T1) and post-intervention (T2; around 3 months after randomisation). Longitudinal cohort assessment (both arms) will take place around 12 months after randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Immediate referral to local budget and debt counselling service and a copy of 'Your child, your money', a financial guidance book for new parents
  Interventions: Behavioral: Healthier Wealthier Families
- Waitlist-control arm (Active Comparator): Immediately given a copy of 'Your child, your money' book, and referral to local budget and debt counselling service after a period of 3 months
  Interventions: Behavioral: Healthier Wealthier Families

INTERVENTIONS:
Behavioral: Healthier Wealthier Families — Budget and debt counselling will involve at least one meeting with a counsellor. Examples of assistance the counsellors can offer include: suggestions on ways to improve a participant's financial situation; checking eligibility and helping to apply for social welfare support; helping to organise finances and develop a budget; and assistance with debt management, threatening letters or harassment by debt collectors, or imminent house eviction. The municipal budget and debt counselling services involved in the trial will receive guidance on how to work preventatively with families, which will align with the content of the 'Your child, your money'. The book covers topics such as planning finances, consumer rights, private insurance, family law, parental leave, pensions, saving, and budgeting.

SUMMARY:
Healthier Wealthier Families is a way of working, where child health nurses ask parents about their financial situation and connect them to a free financial help service, if needed. To test whether it helps families, the investigators will randomly select half of the families who want to take part to go to the service straight away and half around 3 months later. Both groups of parents will receive a book about parenting and finances straight away. The investigators will compare how the groups of parents answer on survey questions about meeting the costs of their children's needs, their financial knowledge, financial control, readiness to change, success on personal finance goals, mental health and financial stigma. The investigators predict that the parents who are offered the financial help service straight away will answer more positively on the survey questions. The investigators will ask all parents the survey questions again around 12 months later to see how they are doing.

DETAILED DESCRIPTION:
The Healthier Wealthier Families (HWF) model implements universal screening for economic hardship into child health services and creates a referral pathway to economic support services. To test this, the investigators will conduct a randomised control trial. A longitudinal follow-up with the cohort will explore whether any effects are maintained in the longer-term. The study hypotheses are that families who have received municipal budget and debt counselling services via the HWF model will report a lower rate of child material and social deprivation. Also, that the intervention arm will report greater financial knowledge, financial control, readiness for change, attainment of personal goals to improve one's financial situation, parental mental health and less financial stigma than the waitlist-control arm

ELIGIBILITY:
Inclusion Criteria:

* Parent / caregiver of at least one child aged 0-5 years
* The family is listed at the participating child health care centre
* Parent / caregiver reports at least one risk factor for economic hardship on specified screening questions
* Parent / caregiver lives within the geographical areas served by the participating financial counselling service
* Parent / caregiver has given informed consent

Exclusion Criteria:

* Parent / caregiver does not understand the recruitment invitation.
* Parent / caregiver is already an active user of a financial counselling service.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Child material and social deprivation (MSD) | 3 months after randomisation
  The European Union (EU) measure of child MSD contains 17 items; 13 child-specific items. Parents are asked to indicate whether or not they have the item. If not, they are asked if it is because they cannot afford it (enforced lack) or for another reason (simple lack). Data are collected at the household level; if one child does not have an item it is assumed that all the children in the household lack that item.

SECONDARY OUTCOMES:
Household income and sources of income | 3 months after randomisation
  Overall self-reported household income on an incremental scale up to the median salary for Sweden, and fixed outgoings (e.g. rent and bills) to calculate the net income for the household. Also, selection of all applicable sources of income from a list, which includes all available benefits in Sweden
Financial knowledge | 3 months after randomisation
  A selection of questions covering financial knowledge and where to turn for help for better control over finances and debt management will be taken from a survey conducted by the Swedish Consumer Agency survey
Financial control | 3 months after randomisation
  A 9-item measure of financial control will be used. Respondents will be asked to indicate the extent to which they agree or disagree with a series of nine statements using a 5-point scale, ranging from 1 (strongly disagree) to 5 (strongly agree).
Readiness for change | 3 months after randomisation
  To assess readiness for change, participants will be asked to complete a Readiness Ruler regarding changing their financial situation. The ruler will employ a 0-10 visual analogue scale. Scores of 1-3 represent non-readiness to change, scores of 4-6 uncertainty, scores of 7-8 represent readiness, and 9-10 represent ongoing attempts at changing.
Personal goal | 3 months after randomisation
  Participants will be asked to write a personal goal for improving their financial situation at T1. Their own words will be presented back to them at T2 and T3, and they will be asked to rate how far they have achieved their goal. A visual analogue scale ranging from anchors "not at all" for the value 0 to "extremely" for the value 10 will be used.
Parental mental health | 3 months after randomisation
  The 12-Item General Health Questionnaire (GHQ-12). Respondents are asked to rate the degree to which they have experienced a symptom during the last week with four response categories (e.g. less than usual, no more than usual, rather more than usual, or much more than usual). The minimum score is 0, and the maximum is 36. A higher score indicates a higher levels of distress.
Perceived financial stigma | 3 months after randomisation
  An 8-item measure of perceived financial stigma will be used. Respondents are asked to indicate the extent to which they agree or disagree with a series of eight statements using a 5-point scale, ranging from 1 (definitely disagree) to 5 (definitely agree).

CONTACTS AND LOCATIONS:
Overall Officials: Anna Sarkadi, Prof, Principal Investigator — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Uppland, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johansson N, Sarkadi A, Isaksson D, Warner G. Feasibility of a randomised controlled trial of Healthier Wealthier Families in Sweden: results from the Ameliorating Child poverty through Connecting Economic Services with child health Services (ACCESS) pilot study. BMC Health Serv Res. 2025 Dec 1;25(1):1561. doi: 10.1186/s12913-025-13753-y. PMID 41327350
- [Derived] Johansson N, Sarkadi A, Feldman I, Price AMH, Goldfeld S, Salonen T, Wijk K, Isaksson D, Kolic E, Stenquist S, Elg M, Lonn E, Wennelin J, Lindstrom L, Medina M, Aberg S, Viklund J, Warner G. Ameliorating Child poverty through Connecting Economic Services with child health Services (ACCESS): study protocol for a randomised controlled trial of the healthier wealthier families model in Sweden. BMC Public Health. 2022 Nov 25;22(1):2181. doi: 10.1186/s12889-022-14424-x. PMID 36434580